CLINICAL TRIAL: NCT07176442
Title: Enhancing Teaching Strategies for Newly Recruited Interns: A Randomized Controlled Trial Comparing Massive Open Online Courses, Simulation, and Escape Games
Brief Title: Enhancing Teaching Strategies for Newly Recruited Interns: Comparing Massive Open Online Courses, Simulation, and Escape Games
Acronym: PEDAGO-INT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed V Souissi University (Other)
Responsible Party: Principal Investigator, Safae Dehbi, Principal Investigator, Mohammed V Souissi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INTERN-PEDAGOGY-TRIAL-2025
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Medical Education
Keywords: Medical Education; Randomized Controlled Trial; E-Learning; Simulation Training; Gamification

STUDY DESIGN:
Intervention Model Description: Fifty-one newly recruited medical interns will be randomly assigned in equal proportions to one of three parallel groups. Each group will receive a single, distinct educational intervention on the same clinical case (diabetic ketoacidosis). The interventions are: (1) a structured MOOC with interactive quizzes, (2) a high-fidelity simulation scenario with debriefing, or (3) a gamified escape game composed of 10 puzzles. Participants remain in their assigned group throughout the study, and outcomes are compared between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MOOC (E-learning) (Experimental): Participants complete a structured Massive Open Online Course (MOOC) hosted on Canvas. The course includes four 4-5 minute video modules on diabetic ketoacidosis, with interactive quizzes between modules.
  Interventions: Behavioral: MOOC (E-Learning)
- Simulation (Experimental): Participants take part in a high-fidelity simulation session using a mannequin programmed for diabetic ketoacidosis management. Each session is followed by a structured debriefing led by the instructor.
  Interventions: Behavioral: Simulation Training
- Escape Game (Experimental): Participants join a 30-minute educational escape game with 10 puzzles that guide them through the diagnosis and management of diabetic ketoacidosis. The activity emphasizes collaboration and problem-solving.
  Interventions: Behavioral: Educational Escape Game

INTERVENTIONS:
Behavioral: MOOC (E-Learning) — Participants complete a structured Massive Open Online Course (MOOC) hosted on Canvas. The course includes four 4-5 minute video modules on diabetic ketoacidosis, with interactive quizzes between modules.
  Arms: MOOC (E-learning)
Behavioral: Simulation Training — Participants take part in a high-fidelity simulation session using a mannequin programmed for diabetic ketoacidosis management. Each session is followed by a structured debriefing led by the instructor.
  Arms: Simulation
Behavioral: Educational Escape Game — Participants join a 30-minute educational escape game with 10 puzzles that guide them through the diagnosis and management of diabetic ketoacidosis. The activity emphasizes collaboration and problem-solving.
  Arms: Escape Game

SUMMARY:
This randomized controlled trial will compare three innovative teaching methods-Massive Open Online Courses (MOOCs), simulation, and escape games-among newly recruited medical interns at Ibn Sina University Hospital in Rabat, Morocco. The study aims to evaluate their effectiveness in improving knowledge of diabetic ketoacidosis management, retention of knowledge after 4 weeks, and learner motivation. Fifty-one interns will be randomly assigned to one of the three groups. Outcomes will be assessed using multiple-choice knowledge tests at baseline, immediately after training, and 4 weeks later, as well as the Intrinsic Motivation Inventory questionnaire. The results will provide evidence on the most effective and engaging approach to support induction training of new medical interns.

DETAILED DESCRIPTION:
The induction period for newly recruited medical interns represents a critical stage in their professional training. On arrival at the hospital, interns must rapidly acquire clinical knowledge, technical skills, and adaptive behaviors to ensure patient safety and integration into the healthcare team. Innovative teaching strategies, including Massive Open Online Courses (MOOCs), high-fidelity simulation, and gamified approaches such as escape games, have been increasingly adopted in medical education, but comparative evidence of their effectiveness in this context remains limited.

This study is a prospective, randomized controlled trial conducted at Ibn Sina University Hospital, Rabat, Morocco. A total of 51 newly recruited medical interns will be randomly assigned to one of three intervention groups:

MOOC group: A structured online course hosted on Canvas, including four short video modules (4-5 minutes each) covering diagnosis, pathophysiology, precipitating factors, and therapeutic management of diabetic ketoacidosis (DKA). Interactive quizzes are included between modules.

Simulation group: Participants engage in a high-fidelity simulation scenario of DKA secondary to urinary tract infection, using a mannequin in a controlled training environment. Each session is followed by a structured debriefing.

Escape game group: Interns participate in a 30-minute collaborative escape game consisting of 10 puzzles designed to guide them through the diagnostic and therapeutic steps of DKA management, encouraging teamwork and problem-solving.

All interventions focus on the same clinical case to ensure content comparability. A single faculty member oversees all sessions to maintain consistency in delivery and evaluation.

Outcomes: Knowledge acquisition is assessed using a validated 10-item multiple-choice questionnaire administered at baseline (pre-test), immediately after the intervention (post-test), and 4 weeks later (late post-test) to evaluate both immediate learning and short-term retention. Motivation and satisfaction are assessed immediately after the intervention using the Intrinsic Motivation Inventory (IMI), focusing on interest/enjoyment, perceived competence, perceived choice, and pressure/tension.

Analysis: Scores will be compared within and between groups using repeated-measures ANOVA and appropriate non-parametric tests. The study is designed to test whether one teaching method provides superior short-term knowledge gains, improved retention, or greater learner motivation.

This trial addresses an important gap in medical education by directly comparing three pedagogical approaches during the induction training of new interns. Results are expected to guide educational policy and support the development of blended learning strategies that combine the strengths of digital, experiential, and gamified methods.

ELIGIBILITY:
Inclusion Criteria:

* Newly recruited medical interns at Ibn Sina University Hospital (CHU), Rabat
* Voluntary participation with signed informed consent
* No prior formal training specifically focused on diabetic ketoacidosis

Exclusion Criteria:

* Refusal to participate
* Previous advanced training on diabetic ketoacidosis management

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Immediat Change in knowledge score on diabetic ketoacidosis (DKA) MCQ | Baseline (pre-test) and immediately after the intervention (same day)
  Ten-item multiple-choice questionnaire (0-10 points) covering DKA diagnosis, severity, triggers, and initial management. Score at post-test minus pre-test; higher values indicate greater knowledge gain. Administered identically across all three arms (MOOC, Simulation, Escape Game) using the same validated items. Safety Issue: No.

SECONDARY OUTCOMES:
Change in knowledge score from baseline to 4-week follow-up | Baseline and 4 weeks after intervention
  Same 10-item MCQ (0-10); follow-up minus baseline. Higher values indicate better retention. Safety Issue: No.
Intrinsic Motivation Inventory (IMI) scores | Immediately after the intervention (same day)
  The IMI is a validated self-report tool based on self-determination theory. In this study, four subscales are assessed on a 7-point Likert scale:
  Interest/Enjoyment (higher scores = greater engagement) Perceived Competence (higher scores = greater self-efficacy) Perceived Choice (higher scores = stronger sense of autonomy) Pressure/Tension (higher scores = greater stress; lower scores desirable). Median scores across groups will be compared to evaluate motivational impact of MOOC, simulation, and escape game interventions. Safety Issue: No.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medecine And Pharmacy Of Rabat, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Issenberg SB, McGaghie WC, Petrusa ER, Lee Gordon D, Scalese RJ. Features and uses of high-fidelity medical simulations that lead to effective learning: a BEME systematic review. Med Teach. 2005 Jan;27(1):10-28. doi: 10.1080/01421590500046924. PMID 16147767
- [Background] Khanna A, Ravindran A, Ewing B, Zinnerstrom K, Grabowski C, Mishra A, Makdissi R. Escape MD: Using an Escape Room as a Gamified Educational and Skill-Building Teaching Tool for Internal Medicine Residents. Cureus. 2021 Sep 27;13(9):e18314. doi: 10.7759/cureus.18314. eCollection 2021 Sep. PMID 34725586
- [Background] Alturkistani A, Lam C, Foley K, Stenfors T, Blum ER, Van Velthoven MH, Meinert E. Massive Open Online Course Evaluation Methods: Systematic Review. J Med Internet Res. 2020 Apr 27;22(4):e13851. doi: 10.2196/13851. PMID 32338618